CLINICAL TRIAL: NCT06700746
Title: Efficacy of Dextrose Prolotherapy Compare With Extracorporeal Shock Wave Therapy in the Treatment of Chronic Rotator Cuff Tendinopathy
Brief Title: Efficacy of Dextrose Prolotherapy Compare With ESWT in the Treatment of Chronic Rotator Cuff Tendinopathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Songsuda Roongsaiwatana, Principal Investigator, Mahidol University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: COA.No.MURA2023/839
Record Dates: First submitted 2024-11-20; First posted 2024-11-22 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Chronic Rotator Cuff Tendinopathy
MeSH Terms: interventions — Prolotherapy; Extracorporeal Shockwave Therapy

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prolotherapy (Experimental): Solution 3.6 mL of 25% dextrose and 0.4 mL xylocaine total 4.0 mL And Solution 3.5 mL of 15% dextrose and 0.8 mL xylocaine total 4.3 mL each site Injection interval week 0, 3 and 6 Ultrasound guided injection Injection into enthesis points
  Interventions: Procedure: Prolotherapy
- Extracorporeal shock wave therapy (ESWT) (Active Comparator): ESWT Treatment interval week 0, 1 and 2 Energy intensity 0.20-0.25 mJ/mm2 per impulse Frequency 4-5 Hz for 2,000 shocks
  Interventions: Device: Extracorporeal shock wave therapy (ESWT)

INTERVENTIONS:
Procedure: Prolotherapy — Prolotherapy is an injection of a relatively small volume of an irritant or sclerosing solution at sites of painful ligament and/or tendon insertions, and in adjacent joint space over the course of several treatment sessions
  Arms: Prolotherapy
Device: Extracorporeal shock wave therapy (ESWT) — Extracorporeal shock wave therapy (ESWT), a kind of physical modalities, generating acoustic pulses, that are high positive pressure amplitudes, subsequently transferring concentrated energy to small focal distant areas of 2-8 mm in diameter
  Arms: Extracorporeal shock wave therapy (ESWT)

SUMMARY:
To compare the efficacy of dextrose solution injection with ESWT for pain reduction in rotator cuff tendinopathy.

Additionally, secondary objective is to evaluate DASH and active range of motion of shoulder joint

ELIGIBILITY:
Inclusion Criteria:

* Chronic shoulder pain for at least 3 months
* Unilateral affected side
* History of unsuccessful conservative treatment
* Age 18 years or older

Exclusion Criteria:

* Rotator cuff complete tear
* Local or generalized arthritis
* Previous shoulder surgery
* Previous history allergy to local anesthesia
* Pregnancy
* Current infectious or tumorous disease
* Dysfunction in the neck or thoracic region of both
* Coagulation disturbance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2023-11-10 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2024-11-20 (Actual)

PRIMARY OUTCOMES:
VAS score | Assessment at baseline, three weeks, six weeks, three months and six months after the end of the treatment
  Pain reduction VAS

SECONDARY OUTCOMES:
Function DASH score | Assessment at baseline, three weeks, six weeks, three months and six months after the end of the treatment
  Disabilities of the arm, shoulder and hand
Shoulder ROM | Assessment at baseline, three weeks, six weeks, three months and six months after the end of the treatment
  Active range of motion:
  Forward flexion Abduction Internal rotation External rotation
  Active range of motion:
  Forward flexion Abduction Internal rotation External rotation
  Active range of motion:
  Forward flexion Abduction Internal rotation External rotation

CONTACTS AND LOCATIONS:
Overall Officials: Songsuda Roongsaiwatana, M.D., Study Director — Ramathibodi Hospital
Locations (1):
- Physical medicine and rehabilitation, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hauser RA, Lackner JB, Steilen-Matias D, Harris DK. A Systematic Review of Dextrose Prolotherapy for Chronic Musculoskeletal Pain. Clin Med Insights Arthritis Musculoskelet Disord. 2016 Jul 7;9:139-59. doi: 10.4137/CMAMD.S39160. eCollection 2016. PMID 27429562
- [Background] Galasso O, Amelio E, Riccelli DA, Gasparini G. Short-term outcomes of extracorporeal shock wave therapy for the treatment of chronic non-calcific tendinopathy of the supraspinatus: a double-blind, randomized, placebo-controlled trial. BMC Musculoskelet Disord. 2012 Jun 6;13:86. doi: 10.1186/1471-2474-13-86. PMID 22672772